CLINICAL TRIAL: NCT05855629
Title: "A Comparative Clinical Evaluation of the Efficacy of Topical Adapalene, Benzoyl Peroxide Gel, Oral Lactobacillus Rhamnosus, D-chiro-inositol, Inulin Capsule, and Their Fixed Combination in Mild to Moderate Acne Vulgaris Patients."
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Treatment and Diagnostic Center of Private Enterprise "Asklepiy" (Other)
Collaborators: delta medical promotions ag (Unknown)
Responsible Party: Principal Investigator, Yuriy Andrashko, Yuriy Andrashko, Treatment and Diagnostic Center of Private Enterprise "Asklepiy"
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDA1370
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Inulin; Adapalene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical Adapalene, Benzoyl Peroxide Gel (Other)
  Interventions: Drug: Topical Adapalene, Benzoyl Peroxide Gel
- Oral Lactobacillus Rhamnosus, D-chiro-inositol, Inulin Capsule (Other)
  Interventions: Dietary Supplement: Oral Lactobacillus Rhamnosus, D-chiro-inositol, Inulin Capsule
- Topical Adapalene,Benzoyl Peroxide Gel,Oral Lactobacillus Rhamnosus,D-chiro-inositol,Inulin Capsule (Other)
  Interventions: Dietary Supplement: Oral Lactobacillus Rhamnosus, D-chiro-inositol, Inulin Capsule; Drug: Topical Adapalene, Benzoyl Peroxide Gel

INTERVENTIONS:
Dietary Supplement: Oral Lactobacillus Rhamnosus, D-chiro-inositol, Inulin Capsule — Lactobacillus Rhamnosus 1,5 х 10*9, Inulin 25mg, D-chiro-inositol 250mg
  Arms: Oral Lactobacillus Rhamnosus, D-chiro-inositol, Inulin Capsule; Topical Adapalene,Benzoyl Peroxide Gel,Oral Lactobacillus Rhamnosus,D-chiro-inositol,Inulin Capsule
Drug: Topical Adapalene, Benzoyl Peroxide Gel — Adapalene 1mg/g, Benzoyl Peroxide 25mg/ml
  Arms: Topical Adapalene, Benzoyl Peroxide Gel; Topical Adapalene,Benzoyl Peroxide Gel,Oral Lactobacillus Rhamnosus,D-chiro-inositol,Inulin Capsule

SUMMARY:
The study aims to conduct a comparative clinical evaluation of the effectiveness of a fixed topical combination of adapalene with benzoyl peroxide in the form of a gel, a fixed combination of Lactobacillus rhamnosus, D-chiro-inositol and inulin in the form of capsules and their combination in patients with acne vulgaris of mild and moderate severity and laboratory lipid analysis profile of sebum, lipid metabolism, and IGF-1 (insulin-like growth factor).

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate level of Acne Vulgaris

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-06-12 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
GAGS (Global Acne Grading System) | 180 days
  The primary end point of the study is the intensity of acne manifestations according to the GAGS scale

SECONDARY OUTCOMES:
IGA (Investigator Global Assessment) | 180 days
  The secondary end point of the study is the intensity of acne manifestations according to the IGA scale

CONTACTS AND LOCATIONS:
Locations (1):
- TDC PE "Asklepiy", Uzhhorod, Zakarpattia Oblast, Ukraine